CLINICAL TRIAL: NCT01408797
Title: A Prospective, Open-Label, Pilot Study of Clonal Deletion on Living-Relative Donor Kidney Transplantation
Brief Title: Clonal Deletion on Living-Relative Donor Kidney Transplantation
Acronym: DAWN
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fuzhou General Hospital (Other)
Collaborators: Terasaki Foundation (Unknown)
Responsible Party: Fuzhou General Hospital, Tan Jianming, MD,PhD
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAWN-2011-TJM
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-02

CONDITIONS: Renal Transplantation; Uremia
Keywords: clonal deletion; kidney transplantation
MeSH Terms: conditions — Uremia | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Donor specific transfusion (Experimental): Subjects with uremia will undergo donor specific transfusion before transplantation
  Interventions: Procedure: donor specific transfusion
- Clonal deletion (Experimental)
  Interventions: Drug: MMF, Bortezomib
- Drugs Added When Needed (Experimental)
  Interventions: Procedure: drugs added according to the immuno condition of the recipients

INTERVENTIONS:
Procedure: donor specific transfusion — before transplantation,200mL of donor whole blood will be transfused to the recipient
  Arms: Donor specific transfusion
Drug: MMF, Bortezomib — MMF and Bortezomib will be administered after donor specific transfusion
  Arms: Clonal deletion
Procedure: drugs added according to the immuno condition of the recipients — drugs (corticosteroid, MMF and/or CNI) will be added according to the recipients immuno event and donor specific antibody
  Arms: Drugs Added When Needed

SUMMARY:
The objective of this trial is to determine if clonal deletion before kidney transplantation can effectively reduce the need for post transplant immunosuppression. The investigators will adapt a DAWN (Drugs (immunosuppressants) Added When Needed) treatment protocol to assess the effect of clonal deletion and closely monitor acute rejection, renal function, and graft survival. 15 patients eligible for the study as described below will be enrolled.

DETAILED DESCRIPTION:
The objective of this trial is to determine if clonal deletion can effectively reduce the need for post transplant immunosuppressive medicine. Emphasis will be placed on adverse events that are associated with clonal deletion. The investigators will assess whether DAWN (Drugs (immunosuppressants) Added When Needed) is feasible in living-relative donor kidney transplantation and the effectiveness of clonal deletion treatment on the rate of rejection, patient survival, and graft function from day 0 to 12 months after transplantation. Numbers of patients on single drug and dual therapy immunosuppression will be counted. Additionally, the investigators would assess time to immune event (rejection or antibody), the severity of acute rejection or antibody mediated rejection by Banff criteria, the incidence of delayed graft function (defined as the need for post-transplant dialysis), and the incidence of adverse events including infection, grade 3 and above non-hematologic toxicities, and grade 4 hematologic toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Uremia patient of any race that is greater than or equal to 18 years of age but less than 60 years old
2. Recipients of a kidney from a certifiable relative donor 18-60 years of age
3. Patient is willing and capable of giving written informed consent for study participation and able to participate in the study for 12 months

Exclusion Criteria:

1. Women who are pregnant, intend to become pregnant in the next 1 years, breastfeeding, or have a positive pregnancy test on enrollment or prior to study medication administration
2. Patient with prior solid organ transplant or cell transplant (e.g. bone marrow or islet cell).
3. Patient is deemed likely to have a second solid organ transplant or cell transplant (e.g. bone marrow or islet cell) in next 3 years
4. Patient receiving a concurrent SOT (heart, liver, pancreas) or cell transplant (islet, bone marrow, stem cell)
5. ABO incompatible donor recipient pair or CDC crossmatch positive transplant
6. Sensitized patients (most recent anti-HLA Class I or II Panel Reactive Antibodies (PRA)>0% by a CDC-assay) or patients identified a high immunological risk by the transplant physician
7. Donor with cardiac death (non-heart beating donor)
8. Recipient CMV seronegative receiving a organ from a seropositive donor (CMV seromismatch)
9. Donor OR Recipient are known hepatitis C antibody-positive or polymerase chain reaction (PCR) positive for hepatitis C
10. Donors OR Recipient are known hepatitis B surface antigen-positive or PCR positive for hepatitis B AND recipient is HBV negative
11. Patient and/or donors with known human immunodeficiency virus (HIV) infection
12. Patient at risk for tuberculosis (TB) Current clinical, radiographic, or laboratory evidence of active or latent TB as determined by local standard of care

    History of active TB:

    Within the last 2 years, even if treated Greater than 2 years ago, unless there is documentation of adequate treatment according to locally accepted clinical practice Patient at risk of reactivation of TB precludes administration of conventional immunosuppression (as determined by investigator and based upon appropriate evaluation)
13. Patient with any significant infection or other contraindication that would preclude transplant
14. Patient with a history of hypercoaguable state
15. Patient with a history of substance abuse (drugs or alcohol) within the past 6 months, or psychotic disorders that are not compatible with adequate study follow-up.
16. Patient with active peptic ulcer disease (PUD), chronic diarrhea, or gastrointestinal malabsorption
17. Patient with a history of cancer within the last 5 years (exception: non-melanoma skin cell cancers cured by local resection are permitted)
18. Patient with a chest radiograph (no more than 2 months prior to randomization) consistent with an acute lung parenchymal process and malignancy
19. Patient with a hypersensitivity to any study drugs
20. Patient who have used any investigational drug within 30 days prior to the Day 1 visit
21. . Patients with autoimmune disease or patient treated with immunosuppressive therapy (eg methotrexate, abatacept, etc) for indications such as autoimmune disease or patient with comorbidity to a degree that treatment with such agents is likely during the trial
22. Prisoner or patient compulsorily detained (involuntarily incarcerated) for treatment or either a psychiatric or physical (e.g. infectious disease) illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Dosage of immunosuppressants | one year
  Effectiveness of clonal deletion on reducing the dosage of immunosuppressants (calcineurin inhibitor plus mycophenolate, azothioprine, or sirolimus).

SECONDARY OUTCOMES:
immune event | 1 year
  Time to immune event (acute rejection or DSA);
DSA | 1 year
  Proportion of patients who become positive for donor specific HLA antibodies post transplant
DGF | 1 years
  Incidence of delayed graft function (defined as need for post-transplant dialysis)
Renal function | 1 year
  Change in renal function as determined by estimated glomerular filtration rate and proteinuria (>1g) at 1 year post transplant
Survival | 1 year
  Allograft Survival at 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Tan Jianming, MD,PhD, Principal Investigator — Fuzhou General Hospital
Locations (1):
- No. 156, Xi er huan Road, Fuzhou, Fujian, China